## Statistical analysis

Official title: Effects of deep neuromuscular block on surgical pleth index-guided remifentanil administration in laparoscopic herniorrhaphy: A prospective randomized trial

NCT number: NCT04022733

**Document date:** Jan 18, 2022

Institution Name: Ajou University School of Medicine

The primary outcome was the infusion rate of remifentanil during pneumoperitoneum. Based on the findings of a previous study, we considered a difference in remifentanil infusion rate >0.032  $\mu$ g/kg/min (16% of mean infusion rate of remifentanil in moderate NMB under SPI-guided anesthesia for laparoscopic surgery [mean infusion rate of 0.192 (SD 0.064)  $\mu$ g/kg/min]) as clinically relevant. Based on a significance level of 5% and statistical power of 80%, each group required 63 subjects for analysis. We enrolled a total of 134 patients to compensate for dropouts and observational variation.

Statistical analyses were conducted using SPSS software version 25.0 (IBM, NY, USA). Data are presented as mean  $\pm$  SD, median (interquartile range), and number of patients. The normality of distribution was tested using the Kolmogorov–Smirnov/ the Shapiro–Wilk test. Continuous data were compared using a two-tailed t test when normally distributed; however, Mann-Whitney *U*-test was used for non-normally distributed data. Categorical data were compared using the Chi-square test or Fisher's exact test, as appropriate. Intergroup comparisons for repetitively measured data were performed by unpaired t-test with Bonferroni correction. *P*-values < 0.05 were considered statistically significant.